CLINICAL TRIAL: NCT02963285
Title: Optimal Positioning of Nasopharyngeal Temperature Probes in Pediatric Patients: A Prospective Cohort Study
Brief Title: Optimal Positioning of Nasopharyngeal Temp Probe
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, John Zhong, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 072016-059
Record Dates: First submitted 2016-11-09; First posted 2016-11-15 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Pediatric Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 0 to 6 months
  Interventions: Other: Nasopharyngeal temperature probe
- 7 months to less than 1 year
  Interventions: Other: Nasopharyngeal temperature probe
- 1 to less than 2 years
  Interventions: Other: Nasopharyngeal temperature probe
- 2 to less than 6 years
  Interventions: Other: Nasopharyngeal temperature probe
- 6 to 12 years
  Interventions: Other: Nasopharyngeal temperature probe

INTERVENTIONS:
Other: Nasopharyngeal temperature probe — Nasopharyngeal temperatures will initially be recorded 30 minutes after induction of anesthesia. Nasopharyngeal probes will then be withdrawn at the designated increment for each age group and will be equilibrated for 3 minutes before the temperature is recorded. Thereafter, the nasopharyngeal withdrawal sequence will be repeated.

SUMMARY:
The purpose of this study is to determine the optimal range of insertion depths for a nasopharyngeal probe in anesthetized pediatric patients as a function of age.

DETAILED DESCRIPTION:
Before surgery, the esophageal and nasopharyngeal probes (DeRoyal GP/Nasopharyngeal Probe, 9F, 400 series [REF 81-025409] to be used in a given patient will be connected to the two channels of the clinical monitor in the designated room. The tips will be inserted at least five centimeters into a well stirred container of water maintained near 370 Celsius. Temperatures will be recorded from each, and the offset (if any) used as a correction factor in the statistical analysis below.

After anesthetic induction and intubation, patients will be positioned per clinical routine for the selected operation. An esophageal temperature probe (DeRoyal General Purpose Temperature Probe, SOFT 9 French, 400 series [REF V81-010400]) will be inserted. The optimal placement of the esophageal temperature probe varies based on the height of the patient8. Broad consensus is that the measurement is most accurate in the distal third of the esophagus. The use of acoustic criteria for optimal placement is not a reliable method9. Bloch et al.,5 proposed the use of a simple formula of one quarter of the patient's height plus 4.5 centimeters with the upper incisors as the starting point. This technique reliably locates the tip of the probe 2 centimeters above the lower esophageal sphincter.

For the two groups of infants aged up to twelve months, the nasopharyngeal probe will be marked with indelible ink from 2-10 cm in 1-cm increments and inserted 10 cm. For the two groups of children between 1 and 5 years, the nasopharyngeal probe will be marked with indelible ink from 2-15 cm in 1.5-cm increments and inserted 15 cm. For older children, a nasopharyngeal probe will be marked with indelible ink from 2 to 20 cm at 2 cm increments from its tip, and inserted 20 cm. In each case, investigators will confirm under direct vision that the probe tip is visible in the oropharynx. Insertion will be repeated if necessary; the contralateral nostril or a new probe can be used.

Both nasopharyngeal and esophageal temperatures will initially be recorded 30 minutes after induction of anesthesia. Nasopharyngeal probes will then be withdrawn at the designated increment for each age group and will be equilibrated for 3 minutes before the temperature is recorded. Thereafter, the nasopharyngeal withdrawal sequence will be repeated. The number of measurement will depend on the initial depth of insertion; with measurements continuing until only 2 centimeters remain in the nostril.

Temperature in the operating room will be maintained per clinical routine. Normothermia will be maintained with forced-air warmer and if necessary with overhead warming lights per clinical routine.

ELIGIBILITY:
Inclusion Criteria:

1. Elective non-cardiac surgery in children to last at least 1.5 hours;
2. Supine position anticipated;
3. General endotracheal anesthesia.

Exclusion Criteria:

1. Nasopharyngeal disease (e.g. sinusitis), upper airway abnormalities, or planned oral or facial surgery;
2. History of genetic or congenital anomalies leading to facial dimorphism;
3. History of recent substantive epistaxis or suspected bleeding disorder;
4. Therapeutic-dose anti-coagulation;
5. Contraindication to esophageal temperature probe insertion (i.e., esophageal varices, congenital anomalies).

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subjects will be pediatric patients having elective non-cardiac surgery with general anesthesia and endotracheal intubation at the Children's Health.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Difference between esophageal temp and nasopharyngeal temp | 5 minute increments at each position
  Nasopharyngeal probe will be withdrawn incrementally, with 5 minutes to equilibrate at each depth.

CONTACTS AND LOCATIONS:
Overall Officials: John Zhong, MD, Principal Investigator — UTSouthwestern Medical Center
Locations (1):
- Children's Health Children's Medical Center Dallas, Dallas, Texas, United States